CLINICAL TRIAL: NCT06181149
Title: Auditory Prediction and Error Evaluation in the Speech of Individuals Who Stutter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Washington (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DC020162 (NIH); 1R01DC020162-01A1 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2023-12-26 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subjects; Stuttering, Developmental
Keywords: stuttering
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental)
  Interventions: Behavioral: Delaying speech initiation
- Group 2 (Experimental)
  Interventions: Behavioral: Auditory errors and pre-speech auditory modulation
- Group 3 (Experimental)
  Interventions: Behavioral: Contributions of the speech premotor cortex to pre-speech auditory modulation
- Group 4 (Experimental)
  Interventions: Behavioral: Delaying auditory feedback

INTERVENTIONS:
Behavioral: Delaying speech initiation — This intervention will examine the effects of misalignment between prediction and auditory feedback in participants. We will use transcranial magnetic stimulation to induce a temporal misalignment between prediction and auditory feedback while participants produce speech.
  Arms: Group 1
Behavioral: Auditory errors and pre-speech auditory modulation — This intervention will examine the contributions of auditory errors to pre-speech auditory modulation. Participants will receive auditory perturbations while speaking, and we will collect their brain activities throughout the study.
  Arms: Group 2
Behavioral: Contributions of the speech premotor cortex to pre-speech auditory modulation — This intervention will examine the effects of stimulation of the left ventral premotor cortex on pre-speech auditory modulation. Participants will receive electrical stimulation while speaking.
  Arms: Group 3
Behavioral: Delaying auditory feedback — This intervention will examine the effects of misalignment between prediction and auditory feedback in participants. We will use delayed auditory feedback to induce a temporal misalignment between prediction and auditory feedback while participants produce speech.
  Arms: Group 4

SUMMARY:
Stuttering negatively impacts communication and reduces the overall quality of life and well-being of individuals who stutter. This study will provide a strong foundation for developing neural and behavioral interventions for stuttering. Participants will be asked to name pictures, read words/sentences silently or aloud, and listen to speech and nonspeech sounds while their speech, muscle, and brain signals are collected. Some participants may also receive brain stimulation while reading and speaking.

ELIGIBILITY:
Inclusion Criteria:

* being a monolingual, native speaker of American English
* absence of developmental, psychological, neurological, or communication disorders (other than developmental stuttering) as confirmed by a certified research SLP
* normal (age-appropriate) binaural pure-tone hearing threshold (0.5-4k Hz; ≤25 dB HL for younger than 70 years, and ≤35 dB HL for older than 70 years)
* not taking any medications that affect the central nervous system
* absence of safety contra-indication for tDCS, TMS and MRI (for adults)
* scoring at the 20th percentile or higher on standardized speech-language tests (for children)

Exclusion Criteria:

-

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity before and during speaking | within each session of the study that may last up to 2 hours
  Participants will hear speech sounds in each trial before speaking or reading words. Participants' brain activity will be recorded while completing the speaking or reading tasks. The investigators will measure how the participant's brain activity in response to the played sounds changes during speaking and reading tasks. For this purpose, the investigators will measure the amplitude of the brain activity (in microvolts; µV) measured using a commercial electroencephalography system. The amplitude (µV) of the brain signals will be examined both before speaking and during speaking at two time points.
change in speech when participants experience auditory errors | within each session of the study that may last up to 2 hours
  In each trial, participants will experience an auditory error while they produce speech (e.g., they may say "head" but hear "had"). The investigators will measure how the participants' speech changes due to auditory errors that they experience in the current trial. For this p[purpose, the investigators will use commercial microphones to record speech signals and then examine the amplitude of the speech in specific frequency ranges (measured in Hertz; Hz). The frequencies (Hz) of speech in trials with auditory errors will be compared with those without auditory errors.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - Univeristy of Washington, Seattle, Washington